CLINICAL TRIAL: NCT02848404
Title: A Study of Therapeutic Efficacy of Categorical Language Fluency Smartphone Game Application in Mild Cognitive Impairment and Mild Alzheimer's Dementia (Baseline Study)
Brief Title: Therapeutic Efficacy of Categorical Language Fluency Smartphone Game Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Seoul National University (Other); Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Ki Woong Kim, Professor, department of neuropsychiatry, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0028631
Record Dates: First submitted 2016-07-20; First posted 2016-07-28 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Mild cognitive impairment; Cognitive rehabilitation; Cognitive therapy; Alzheimer's disease; Memory enhancement; Categorical language fluency
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Categorical Language Fluency Smartphone Application (Experimental): Smartphone game application specifically aimed at training categorical language fluency
  Interventions: Device: Categorical Language Fluency Smartphone Application

INTERVENTIONS:
Device: Categorical Language Fluency Smartphone Application — 4 weeks' training

SUMMARY:
The purpose of this study is to examine therapeutic efficacy of categorical language fluency smartphone game application in mild cognitive impairment and mild Alzheimer's dementia.

DETAILED DESCRIPTION:
The Categorical Language Fluency Smartphone Game Application was developed based on the semantic distance training, which was effective in improving categorical language fluency of mild cognitive impairment and mild Alzheimer's dementia. 10 patients with mild cognitive impairment and another 10 patients with mild Alzheimer's dementia were recruited to examine therapeutic efficacy of the application.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 55
* Confirmed literacy

  * Diagnosed to mild cognitive impairment by International Working Group on Mild Cognitive Impairment and Clinical Dementia Rating(CDR) of 0 or 0.5.
  * Diagnosed to possible or probable Alzheimer's dementia by NINCDS-ADRDA and Clinical Dementia Rating(CDR) of 1 or below.

Exclusion Criteria:

* Evidence of delirium, confusion
* Any neurological conditions causing cognitive decline such as Parkinson's disease, brain hemorrhage, brain tumor, normal pressure hydrocephalus
* Evidence of severe cerebrovascular pathology
* History of loss-of-consciousness over 1 hour due to head trauma or repetitive head trauma of mild severity
* History of substance abuse or dependence such as alcohol
* Presence of depressive symptoms that could influence cognitive function
* Presence of medical comorbidities that could result in cognitive decline

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Application usage log | 4-weeks treatment
  Log to assess compliance of participant(by describing frequency and duration of training by using application)

SECONDARY OUTCOMES:
Subjective Memory Complaint Questionnaire | after 4-weeks treatment
  to evaluate efficacy of application
Geriatric Depression Scale | after 4-weeks treatment
  to evaluate efficacy of application
Korean version of MMSE for dementia screening | after 4-weeks treatment
  to evaluate efficacy of application

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital, Seong-nam, Korea